CLINICAL TRIAL: NCT00544999
Title: Phase I Study Evaluating the Chemosensitizing Effect of Everolimus Administered With Cytarabine and Daunorubicin in Patients With Acute Myeloid Leukemia in Relapse
Brief Title: Everolimus, Cytarabine, and Daunorubicin in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Recherche Clinique sur les Cancers et le Sang (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000564068; IRLMS-GOELAMS-RAD001; INCA-RECF0476
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Congenital Abnormalities | interventions — Cytarabine; Daunorubicin; Everolimus

INTERVENTIONS:
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: everolimus
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine and daunorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Everolimus may help cytarabine and daunorubicin work better by making cancer cells more sensitive to chemotherapy. Giving everolimus together with cytarabine and daunorubicin may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with cytarabine and daunorubicin in treating patients with relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of everolimus.
* Determine the toxicity of this regimen.

Secondary

* Assess the activation of PI3K/AKT and mTORC 1 in leukemic blasts.
* Evaluate the pharmacokinetics of everolimus at different concentrations.

OUTLINE: This is a multicenter study.

Patients receive primary induction therapy comprising daunorubicin hydrochloride IV on days 1-3, cytarabine IV over 24 hours on day 1, and oral everolimus on days 1 and 7. Patients with more than 5% blasts on day 15 receive a second induction course comprising daunorubicin hydrochloride IV on days 17 and 18 and cytarabine IV twice daily on days 17-20.

After completion of study therapy, patients are followed for 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of de novo or secondary acute myeloid leukemia meeting the following criterion:

  * Relapse > 1 year after obtaining complete remission (any prior treatment allowed)

Exclusion criteria:

* Philadelphia chromosome-positive disease in blast crisis
* FAB M3, M6, or M7 disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Life expectancy ≥ 4 weeks
* Transaminases ≤ 5 times normal
* Creatinine ≤ 2 times normal
* Bilirubin ≤ 3 times normal (except if visceral involvement present)
* Alkaline phosphatase or gamma-glutamyltransferase ≤ 5 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients of must use effective contraception during and for ≥ 28 days after completion of study therapy

Exclusion criteria:

* FEV1 < 30%
* Active uncontrolled or viral pulmonary infection
* Serious psychiatric disorders not related to leukemia or any condition that would prohibit comprehension of the study
* HIV-positive
* Other concurrent malignancy except noninvasive skin cancer or carcinoma in situ
* Patients who are incarcerated or under supervision or trusteeship

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics

Exclusion criteria:

* Prior experimental medication within the past 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of everolimus
Toxicity

SECONDARY OUTCOMES:
Activation of PI3K/AKT and mTORC 1 in leukemic blasts
Pharmacokinetics of everolimus

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Park, MD — Institut de Recherche Clinique sur les Cancers et le Sang
Locations (1):
- Hopital Cochin, Paris, France